CLINICAL TRIAL: NCT06879327
Title: A Phase 2b Multicenter Randomized, Placebo-Controlled, Double-Blind, Study to Evaluate the Safety, Immunogenicity and Efficacy of R21/Matrix-M Malaria Vaccine in African Infants With Different Immunization Schedules
Brief Title: Infant Malaria Vaccine Schedule Optimization
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Serum Institute of India PVT LTD (SII) (Unknown); Agilis (Unknown); Pharmassist Ltd (Industry); MCT-CRO (Unknown); Cytespace (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVIA 108
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Malaria Vaccines
Keywords: Plasmodium falciparum; R21/Matrix-M Malaria Vaccine
MeSH Terms: conditions — Malaria, Falciparum | interventions — Malaria Vaccines; Vaccines, Combined; Vaccines; Rubella Vaccine; MenAfriVac; Yellow Fever Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: 1200 healthy participants will be randomized to an immunization schedule cohort if eligibility is confirmed by the investigator(s) at 42 to 49 days of age. The investigators and parent/legal guardian will both know which immunization schedule cohort their infant has been assigned to.
  Infants will be randomized within each immunization schedule category to a group assignment to either receive the R21/MM or placebo; neither the blinded study staff nor the parent/legal guardian will know whether the infant will receive the R21/MM or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Compressed 6-10-14 Week Schedule: R21/MM Malaria Vaccine (Experimental): Participants will receive R21/MM malaria vaccination at 6, 10, and 14 weeks of age, co-administered with hexavalent vaccine, pneumococcal conjugate vaccine (PCV), and oral rotavirus vaccine (RV). At 9 months of age participants will receive measles-rubella (MR) vaccine, yellow fever (YF) vaccine, and typhoid conjugate vaccine (TCV).
  Participants will receive a booster dose of R21/MM malaria vaccine at 15 months of age co-administered with the 2nd dose of measles-rubella vaccine and meningococcal A conjugate vaccine (MenA).
  Interventions: Biological: R21 Matrix-M (R21/MM) Malaria Vaccine; Biological: Hexavalent Vaccine; Biological: Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Rotavirus, Live Attenuated (Oral) Vaccine; Biological: Measles and Rubella Vaccine; Biological: Meningococcal A conjugate vaccine; Biological: Yellow Fever vaccine; Biological: Typhoid Conjugate vaccine
- Compressed 6-10-14 Week Schedule: Placebo (Placebo Comparator): Participants will receive placebo at 6, 10, and 14 weeks of age, co-administered with hexavalent vaccine, PCV, and oral RV. At 9 months of age participants will receive MR and YF vaccines, and TCV.
  Participants will receive a booster dose of placebo at 15 months of age co-administered with the 2nd dose of MR vaccine and MenA vaccine.
  Participants will receive R21/MM malaria vaccination at 27, 28, and 29 months of age (after completion of the study).
  Interventions: Biological: Placebo; Biological: Hexavalent Vaccine; Biological: Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Rotavirus, Live Attenuated (Oral) Vaccine; Biological: Measles and Rubella Vaccine; Biological: Meningococcal A conjugate vaccine; Biological: Yellow Fever vaccine; Biological: Typhoid Conjugate vaccine
- Relaxed 2-4-6 Month Schedule: R21/MM Malaria Vaccine (Experimental): Participants will receive R21/MM malaria vaccination at 2, 4, and 6 months of age co-administered with hexavalent vaccine, PCV, and oral RV. At 9 months of age participants will receive MR and YF vaccines and TCV.
  Participants will receive a booster dose of R21/MM malaria vaccine at 15 months of age co-administered with the 2nd dose of MR vaccine and MenA vaccine.
  Interventions: Biological: R21 Matrix-M (R21/MM) Malaria Vaccine; Biological: Hexavalent Vaccine; Biological: Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Rotavirus, Live Attenuated (Oral) Vaccine; Biological: Measles and Rubella Vaccine; Biological: Meningococcal A conjugate vaccine; Biological: Yellow Fever vaccine; Biological: Typhoid Conjugate vaccine
- Relaxed 2-4-6 Month Schedule: Placebo (Placebo Comparator): Participants will receive placebo at 2, 4, and 6 months of age co-administered with hexavalent vaccine, PCV, and oral RV. At 9 months of age participants will receive MR and YF vaccines, and TCV.
  Participants will receive a booster dose of placebo at 15 months of age co-administered with the 2nd dose of MR vaccine and MenA vaccine.
  Participants will receive R21/MM malaria vaccination at 27, 28, and 29 months of age (after completion of the study).
  Interventions: Biological: Placebo; Biological: Hexavalent Vaccine; Biological: Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Rotavirus, Live Attenuated (Oral) Vaccine; Biological: Measles and Rubella Vaccine; Biological: Meningococcal A conjugate vaccine; Biological: Yellow Fever vaccine; Biological: Typhoid Conjugate vaccine
- Relaxed 3-6-9 Month Schedule: R21/MM Malaria Vaccine (Experimental): Participants will receive R21/MM malaria vaccination at 3, 6, and 9 months of age. Participants will receive the hexavalent vaccine, PCV, and oral RV at 6 weeks, 10 weeks, and 3 months of age. At 9 months of age participants will receive MR and YF vaccines and TCV.
  Participants will receive a booster dose of R21/MM malaria vaccine at 15 months of age co-administered with the 2nd dose of MR vaccine and the MenA vaccine.
  Interventions: Biological: R21 Matrix-M (R21/MM) Malaria Vaccine; Biological: Hexavalent Vaccine; Biological: Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Rotavirus, Live Attenuated (Oral) Vaccine; Biological: Measles and Rubella Vaccine; Biological: Meningococcal A conjugate vaccine; Biological: Yellow Fever vaccine; Biological: Typhoid Conjugate vaccine
- Relaxed 3-6-9 Month Schedule: Placebo (Placebo Comparator): Participants will receive placebo at 3, 6, and 9 months of age. Participants will receive the hexavalent vaccine, PCV, and oral RV at 6 weeks, 10 weeks, and 3 months of age. At 9 months of age participants will receive MR and YF vaccines and TCV.
  Participants will receive a booster dose of placebo at 15 months of age co-administered with the 2nd dose of MR vaccine and the MenA vaccine.
  Participants will receive R21/MM malaria vaccination at 27, 28, and 29 months of age (after completion of the study).
  Interventions: Biological: Placebo; Biological: Hexavalent Vaccine; Biological: Pneumococcal Polysaccharide Conjugate Vaccine; Biological: Rotavirus, Live Attenuated (Oral) Vaccine; Biological: Measles and Rubella Vaccine; Biological: Meningococcal A conjugate vaccine; Biological: Yellow Fever vaccine; Biological: Typhoid Conjugate vaccine

INTERVENTIONS:
Biological: R21 Matrix-M (R21/MM) Malaria Vaccine — Administered by intramuscular injection. Each 0.5 mL dose contains R21 Malaria Antigen (5 mcg) and Matrix-M1 (Adjuvant) (50 mcg).
  Arms: Compressed 6-10-14 Week Schedule: R21/MM Malaria Vaccine; Relaxed 2-4-6 Month Schedule: R21/MM Malaria Vaccine; Relaxed 3-6-9 Month Schedule: R21/MM Malaria Vaccine
Biological: Placebo — Administered by intramuscular injection. Each dose (0.5 mL) contains Normal saline (0.9%).
  Arms: Compressed 6-10-14 Week Schedule: Placebo; Relaxed 2-4-6 Month Schedule: Placebo; Relaxed 3-6-9 Month Schedule: Placebo
Biological: Hexavalent Vaccine — Administered by intramuscular injection. Each dose of 0.5 mL contains:
  * Diphtheria Toxoid > 30 IU
  * Tetanus Toxoid > 40 IU
  * B. pertussis (whole cell) > 4 IU
  * Hepatitis B surface antigen (HBsAg) (recombinant DNA) 15 mcg
  * Inactivated polio vaccine (Salk strains grown on vero cells): Type - 1 (Mahoney strain) 40 D antigen units (DU); Type - 2 (MEF-1 strain) 8 DU; Type - 3 (Saukett strain) 32 DU
  * Haemophilus influenzae Type b (Hib) Conjugate Vaccine (Adsorbed) polyribosylribitol phosphate (PRP) 10 mcg conjugated to tetanus toxoid (TT) (carrier protein) 19 to 33 mcg]
  Other Names: HEXASIIL
Biological: Pneumococcal Polysaccharide Conjugate Vaccine — Administered by intramuscular injection. Each 0.5 mL dose contains 2 mcg each Saccharide for serotypes 1, 5, 9V, 14, 19A, 19F, 23F, 7F, 6A and 4 mcg Saccharide for serotype 6B.
  Other Names: PNEUMOSIL
Biological: Rotavirus, Live Attenuated (Oral) Vaccine — Administered orally. Each 2.0 mL dose contains: Live Attenuated Bovine-Human Rotavirus Reassortant [G1, G2, G3, G4 and G9], 5.6 focus-forming units (FFU) / serotype.
  Other Names: ROTASIIL
Biological: Measles and Rubella Vaccine — Administered by subcutaneous injection. Each 0.5 mL dose contains not less than 1000 cell culture infectious dose 50% (CCID50) of Measles virus and 1000 CCID50 of Rubella virus.
Biological: Meningococcal A conjugate vaccine — Administered by intramuscular injection. Each 0.5 mL dose contains Meningococcal A polysaccharide 10 mcg and tetanus toxoid (TT) (carrier protein) 10 to 33 mcg.
  Other Names: MenAfriVac
Biological: Yellow Fever vaccine — Yellow fever vaccine will be locally sourced by each trial site in accordance with the countries' EPI program.
Biological: Typhoid Conjugate vaccine — Typhoid conjugate vaccine will be locally sourced by each trial site in accordance with the countries' EPI program.

SUMMARY:
The aim of this study is to identify an optimal infant vaccine schedule for a malaria vaccine which is better aligned with the timing of other vaccine interventions.

DETAILED DESCRIPTION:
The R21/Matrix-M (R21/MM) vaccine has been recommended by the World Health Organization (WHO) to prevent clinical malaria in young children living in moderate to high transmission areas of Sub-Saharan Africa. R21/MM is based on the circumsporozoite protein (CSP) targeting the pre-erythrocytic stage of Plasmodium falciparum. R21/MM elicits high levels of antibodies against the central repeat (Asn-Ala-Asn-Pro [NANP]) of the circumsporozoite protein (CSP) which has been shown to correlate with protection. Currently, R21/MM is recommended to be delivered to young children starting at 5-6 months of age with 3 doses given at monthly intervals, however, there are no existing Essential Programme on Immunization (EPI) vaccine visits scheduled at these ages.

We plan to evaluate, using the R21/MM malaria vaccine as a model system, how age at first vaccine dose and time intervals between doses modify the immunogenicity of the vaccine and the ensuant efficacy in protecting infants against clinical Plasmodium falciparum malaria.

Healthy male or female infants 6 to 7 weeks of age will be randomized to one of three different immunization schedule cohorts: a) a "compressed" conventional schedule at 6-10-14 weeks of age; b) a "relaxed" schedule at 2-4-6 months of age; c) a "relaxed" schedule at 3-6-9 months of age. Participants in each immunization schedule cohort will be randomized in a ratio of 3:1 to receive 4 doses of either R21/MM or placebo with a 4th dose to be administered at 15 months of age.

Infants randomized to the respective immunization schedule categories will receive co-administered routine EPI vaccines. The study will include the provision of a three dose R21/MM compressed schedule to all participants randomized to the placebo arms upon completion of the study at Month 27 of life.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent or thumb-printed and witnessed informed consent obtained from the parent/legal guardian of the infant.
* Infants must have been born full-term (at ≥37 weeks of gestation) and > 2500 grams at birth.
* Immunization schedule Cohorts 1, 2, and 3: : Male and female infants 42-49 days (inclusive) of age at time of enrollment. For infants in Cohort 1, randomization to receive vaccine dose 1 (Groups 1 and 2 of R21/MM or placebo, respectively) will occur at 42-49 days of age. For infants in Cohort 2, randomization to receive vaccine dose 1 (Groups 3 and 4 of R21/MM or placebo, respectively) will occur at 2 months (56-63 days of age). For infants in Cohort 3, randomization to receive vaccine dose 1 (Groups 5 and 6 of R21/MM or placebo, respectively) will occur at 3 months (84-91 days of age).
* The participant's parent/guardian must be willing to avoid travel, particularly in the 28 days after each study vaccination, must confirm willingness to contact the study team in the event of unexpected/unavoidable travel and, for the safety cohort, must confirm availability for the home visits to be conducted by a field worker to collect solicited AEs over the 7 days (day of vaccination and 6 subsequent days) following each study vaccine.
* The participant's parent/guardian must confirm willingness to bring their child to the study clinic / local health care clinic, and capacity to contact the study team in the event the subject has any illnesses or other health concerns during the study.
* Participants who the investigator believes that their parent/guardian can and will comply with the requirements of the protocol (e.g. return for follow-up visits) may be enrolled in the study.

Exclusion Criteria:

* Acute disease at the time of enrolment (acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to participants with a minor illness such as diarrhea, mild upper respiratory infection, without low-grade febrile illness, i.e. axillary temperature < 37.5°C).
* Clinically significant pulmonary, cardiovascular, gastrointestinal, endocrine, neurological, skin, hepatic or renal functional abnormality, as determined by medical history, physical examination or laboratory tests which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial.
* At time of enrollment, any infant who has received any dose of the hexavalent/pentavalent vaccines, pneumococcal vaccine, rotavirus vaccine, IPV or has received more than one dose of oral polio virus or more than one dose of hepatitis B vaccine.
* Weight-for-height/length Z score of less than -3 or other clinical signs of malnutrition.
* Infant with major congenital defects.
* The infant has anaemia associated with clinical signs of symptoms of decompensation, or a haemoglobin of ≤ 5.0 g/dL.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient state (including HIV or asplenia) or known maternal HIV infection (no HIV testing will be routinely done by the study team).
* Administration of immunoglobulins and/or any blood products/blood transfusion from birth to time of planned administration of the vaccine candidate.
* Previous vaccination of participant or biological mother with a malaria vaccine.
* Participation in another research study involving receipt of an investigational product or planned use during the study period.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 42 Days to 49 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2028-03-22 (Estimated); Study Completion 2028-03-22 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMTs) of Anti-circumsporozoite (CS) Immunoglobulin G (IgG) at Baseline and 28 Days after 3rd Vaccine Dose | Baseline and 28 days after 3rd vaccine dose
Geometric Mean Fold Rise (GMFR) in Anti-CS IgG 28 Days after 3rd Vaccine Dose Compared to Baseline | Baseline and 28 days after 3rd vaccine dose
Number of Participants with Solicited Adverse Events | 7 days after each study vaccination
  Local (redness, swelling, and pain at the injection site) and systemic (fever, drowsiness, irritability, decreased appetite) reactions will be collected in a subset of participants (the first 40 participants in each immunization schedule category at each site).
Number of Participants with Unsolicited Adverse Events | 28 days after each study vaccination
Number of Participants with Serious Adverse Events | Up to 27 months of age
Number of Participants with Adverse Events of Special Interest | Up to 27 months of age

SECONDARY OUTCOMES:
Geometric Mean Titers (GMTs) of Anti-CS IgG Before and 28 Days After 4th Vaccine Dose | Month 15 predose and 28 days after vaccination
Fold Increase in Anti-CS IgG Titer Post 4th Dose Compared to Pre-4th Dose | Month 15 predose and 28 days after 4th dose
Number of Clinical Malaria Episodes per Person-year Meeting the Primary Case Definition up to 27 Months | From 6 weeks of age to 27 months of age
  The primary case definition will be P. falciparum asexual parasitemia > 5000 parasites/µL detected by blood slide reading AND presence of fever (axillary temperature ≥ 37.5°C or tympanic temperature ≥ 38°C) or history of fever within 48 hours of presentation at the time of presentation AND occurring in an infant/child who is unwell and brought for treatment to a healthcare facility.
Number of Clinical Malaria Episodes per Person-year Meeting the Primary Case Definition up to 15 Months | From 6 weeks of age to 15 months of age
  The primary case definition will be P. falciparum asexual parasitemia > 5000 parasites/µL detected by blood slide reading AND presence of fever (axillary temperature ≥ 37.5°C or tympanic temperature ≥ 38°C) or history of fever within 48 hours of presentation at the time of presentation AND occurring in an infant/child who is unwell and brought for treatment to a healthcare facility.
Number of Clinical Malaria Episodes per Person-year Meeting the Primary Case Definition from 15.5 to 27 Months | From 15.5 months (2 weeks after the 4th vaccination) to 27 months of age
  The primary case definition will be P. falciparum asexual parasitemia > 5000 parasites/µL detected by blood slide reading AND presence of fever (axillary temperature ≥ 37.5°C or tympanic temperature ≥ 38°C) or history of fever within 48 hours of presentation at the time of presentation AND occurring in an infant/child who is unwell and brought for treatment to a healthcare facility.
Number of Clinical Malaria Episodes per Person-year Meeting the Secondary Case Definition up to 27 Months | From 6 weeks of age to 27 months of age
  The secondary case definition will be P. falciparum asexual parasitemia > 0 parasites/µL detected by blood slide reading and presence of fever (axillary temperature ≥ 37.5°C or tympanic temperature ≥ 38°C) or history of fever within 48 hours of presentation AND occurring in an infant/child who is unwell and brought for treatment to a healthcare facility.
Number of Clinical Malaria Episodes per Person-year Meeting the Secondary Case Definition up to 15 Months | From 6 weeks of age to 15 months of age
  The secondary case definition will be P. falciparum asexual parasitemia > 0 parasites/µL detected by blood slide reading and presence of fever (axillary temperature ≥ 37.5°C or tympanic temperature ≥ 38°C) or history of fever within 48 hours of presentation AND occurring in an infant/child who is unwell and brought for treatment to a healthcare facility.
Number of Clinical Malaria Episodes per Person-year Meeting the Secondary Case Definition from 15.5 to 27 Months | From 15.5 months (2 weeks after the 4th vaccination) to 27 months of age
  The secondary case definition will be P. falciparum asexual parasitemia > 0 parasites/µL detected by blood slide reading and presence of fever (axillary temperature ≥ 37.5°C or tympanic temperature ≥ 38°C) or history of fever within 48 hours of presentation AND occurring in an infant/child who is unwell and brought for treatment to a healthcare facility.

CONTACTS AND LOCATIONS:
Locations (2):
- Burkina Faso (2):
  - Institut de Recherche en Science de la Santé (IRSS), Bobo-Dioulasso
  - Groupe de Recherche Action en Santé (GRAS), Ouagadougou

IPD SHARING:
Plan to Share IPD: Yes
PATH as the Sponsor of the Clinical Study will post the Clinical Trial Data in compliance with the Gates Foundation's Open Access policy and the WHO Joint Statement on Clinical Transparency. The Clinical Trial Data will contain no personally identifiable information (PII) and will be fully anonymized and de-identified.